CLINICAL TRIAL: NCT03869125
Title: Masked Hypertension Evaluated by Automated Office Blood Pressure Measurement (AOBPM) and Office Blood Pressure Measurement (OBPM) in Patients With Obstructive Sleep Apnoea
Brief Title: Masked Hypertension in Patients With Obstructive Sleep Apnoea
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Milan Sova, Head of Sleep Laboratory, Department of Respiratory Medicine, University Hospital Olomouc
Other Study IDs: OSAS_MH
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive sleep apnoea group: Blood pressure measurement
  Interventions: Diagnostic Test: Blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Blood pressure measurement — Blood pressure monitoring using automated office blood pressure measurement (AOBPM), office blood pressure measurement (OBPM), and 24-hour ambulatory blood pressure monitoring

SUMMARY:
Assessment of the possible difference in masked hypertension prevalence when it is evaluated by automated office blood pressure measurement (AOBPM) instead of office blood pressure measurement (OBPM) in patients with obstructive sleep apnoea.

DETAILED DESCRIPTION:
Rationale:

Obstructive sleep apnoea is characterized by repetitive closure of upper airways leading to apnoea (complete airflow cessation) or hypopnoea (airflow limitation > 50%+ blood oxygen desaturation > 4%). It is considered to be an important risk factor for arterial hypertension. In these patients is highly prevalent nocturnal hypertension (NH) and also masked hypertension (MH). Ambulatory blood pressure monitoring (ABPM) is considered to be a gold standard for the diagnosis of NH and MH. Results of ABPM are compared with office blood pressure measurement which could be falsely elevated in some patients (white coat effect). For this reason, automatic office blood pressure measurement was developed. Nowadays some devices like BpTRU were developed. This was validated on some patient groups but robust data for patients with obstructive sleep apnoea are missing.

Process:

Patient with ronchopathy and suspected obstructive sleep apnoea undergo automated office blood pressure monitoring followed by office blood pressure monitoring at the Department of Exercise Medicine and Cardiovascular Rehabilitation. After education, ambulatory blood pressure monitor will be provided to patients for the following 24 hours. In the same night, respiratory polygraphy will be performed in the Sleep Laboratory, Department of Respiratory Medicine, University Hospital Olomouc. All data will be statistically evaluated after completion of the target number of subjects. Patients without obstructive sleep apnoea (apnoea-hypopnoea index < 5) will not be included in statistical evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnoea syndrome

Exclusion Criteria:

* Non- compliance of patients with blood pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected obstructive sleep apnoea syndrome
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
The difference in masked hypertension prevalence between definition I and definition II | 1 day
  Masked hypertension- definition I- office blood pressure measurement < 140/90 mmHg and daytime ambulatory blood pressure measurement > 135/85 mmHg
  Masked hypertension- definition II- automated office blood pressure measurement < 140/90 and daytime ambulatory blood pressure measurement > 135/85 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sova, MD.Ph.D., Principal Investigator — University Hospital Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided